CLINICAL TRIAL: NCT05860738
Title: The Effect of Autoclave Cycles on the Mechanical Properties and Surface Roughness of NITI Archwires: Invivo Study.
Brief Title: The Effect of Autoclave Cycles on the Mechanical Properties and Surface Roughness of NITI Archwires
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Aboalnaga, principal investigator, Cairo University
Other Study IDs: CEBD-CU-2023-5-6
Record Dates: First submitted 2023-05-06; First posted 2023-05-16 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Not Determined
Keywords: surface roughness; modulus of elasticity; NITI archwires; Autoclave cycle
MeSH Terms: interventions — Sterilization

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- As-received NITI archwires: The first group of wires will be investigated in the as-received form (as received from the company without being used clinically).
- Rapid cycle autoclaved NITI archwires: The second group of archwires will be will be installed in the patients mouth for 4 weeks, and then retrieved, cleaned using ultrasonic cleaner, dried and packaged and finally autoclaved using the rapid cycle (4 mins, 134oC)
  Interventions: Other: sterilization
- Universal cycle autoclaved NITI archwires: the third group will be installed in the patients mouth for 4 weeks, and then retrieved, cleaned using ultrasonic cleaner, dried and packaged, the finally autoclaved using the universal cycle (20 mins, 121 oC)
  Interventions: Other: sterilization

INTERVENTIONS:
Other: sterilization — autoclaving using the rapid cycle (4 mins, 134 oC) and the universal cycle (20 mins, 121 oC). The autoclave used in this study is (Anthos A-17 Autoclave, Italy).
  Groups: Rapid cycle autoclaved NITI archwires; Universal cycle autoclaved NITI archwires

SUMMARY:
The aim of this study is to evaluate the effect of different autoclave cycles (universal and rapid cycles) on the surface roughness and mechanical properties of NiTi archwires.

DETAILED DESCRIPTION:
Three groups of 0.016 x 0.022 inch NiTi archwires (American Orthodontics, Wisconsin, USA) will be investigated in this study. The first group of wires will be investigated in the as-received form. The two other groups will be installed in the patients mouth for 4 weeks, and then retrieved, cleaned using ultrasonic cleaner, dried and packaged. The second group will be autoclaved through the rapid cycle (4 mins, 134oC) and the third group will be autoclaved through the universal cycle (20 mins, 121 oC). The autoclave used in this study is (Anthos A-17 Autoclave, Italy).

Each wire will be cut into 3 segments; 2 straight distal segment and one anterior curved segment. The distal segments will be used for tensile testing to derive the mechanical properties and the anterior segment will be used to measure the surface roughness.

The mechanical properties (load deflection curve) will be measured with a universal testing machine (Model 4466, Instron Corp, Canton, Mass) with a 1000-kg load cell at 37°C. Each wire segment will be placed in the jaws of the machine. A grip is positioned at each end of the wire with a distance of 40 mm between the jaws. The machine will be operated in the tensile mode with a crosshead speed of 5 mm per minute. Three characteristics of each sample will be quantified from the readouts: ultimate tensile strength (kg/mm2), elongation rate (%), and modulus of elasticity (kg/mm2).

Atomic force microscopy (AFM) is a non-invasive method for three dimensional analysis of surface roughness. Anterior archwire segments will be evaluated using the AFM (Anton Paar GmbH-Tosca200 AFM, Germany) employing the tapping mode 500 micrometer increment with a rate of 1 line per second. Average surface roughness (Sa) in nanometers will be obtained by software analysis (Mountains 8.2 Software-Digital Surf, Besancon, France). The average surface roughness of each specimen will be measured at three different sites and the mean (Sa) will then be calculated.

ELIGIBILITY:
Inclusion Criteria:

* patients with moderate crowding requiring leveling and alignment

Exclusion Criteria:

* severe crowding.
* extraction cases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: orthodontic patients
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
modulus of elasticity | one month
  springiness of the archwires

SECONDARY OUTCOMES:
surface roughness | one month
  surface roughness of the archwires

CONTACTS AND LOCATIONS:
Locations (1):
- Amira Aboalnaga, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided